CLINICAL TRIAL: NCT01521676
Title: Research of Predictive Clinical and Biological Parameters in Breast Cancer
Brief Title: Predictive Clinical and Biological Parameters in Breast Cancer
Acronym: BC-BIO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BC-BIO/IPC 2009-005
Record Dates: First submitted 2011-12-22; First posted 2012-01-31 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-09

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- breast cancer (Experimental): blood and tumor sample
  Interventions: Genetic: molecular alteration

INTERVENTIONS:
Genetic: molecular alteration — research of molecular alteration

SUMMARY:
Research of predictive clinical and biological factors in breast cancer :

genomic, proteomic, mutation

ELIGIBILITY:
Inclusion Criteria:

* breast cancer
* age > 18
* signed informed consent

Exclusion Criteria:

* emergency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2010-12; Primary Completion 2019-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
molecular alteration in breast cancer | average of 4 weeks after diagnosis
  gene expression level

SECONDARY OUTCOMES:
relation between molecular alteration and clinical and histological characteristics | up to 3 years
  hazard ratio between molecular alteration and clinical and histological characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Carole TARPIN, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (2):
- France (2):
  - Institut Paoli Calmettes, Marseille
  - Hôpital Sainte-Musse, Toulon

REFERENCES:
- [Derived] Goncalves A, Bertucci F, Guille A, Garnier S, Adelaide J, Carbuccia N, Cabaud O, Finetti P, Brunelle S, Piana G, Tomassin-Piana J, Paciencia M, Lambaudie E, Popovici C, Sabatier R, Tarpin C, Provansal M, Extra JM, Eisinger F, Sobol H, Viens P, Lopez M, Ginestier C, Charafe-Jauffret E, Chaffanet M, Birnbaum D. Targeted NGS, array-CGH, and patient-derived tumor xenografts for precision medicine in advanced breast cancer: a single-center prospective study. Oncotarget. 2016 Nov 29;7(48):79428-79441. doi: 10.18632/oncotarget.12714. PMID 27765906
- See also: official web site of the sponsor — http://www.institutpaolicalmettes.fr